CLINICAL TRIAL: NCT00970450
Title: The Central Analgesic Effects of Paracetamol on Serotonergic Pathways
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DAAnaBaselParacetamol 2
Record Dates: First submitted 2009-08-20; First posted 2009-09-02 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Analgesia
Keywords: Paracetamol; Tropisetron; Central analgesic effect; Area of allodynia; Secondary hyperalgesia
MeSH Terms: conditions — Agnosia; Hyperalgesia | interventions — Acetaminophen; Tropisetron

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Paracetamol (Experimental)
  Interventions: Drug: Paracetamol
- Paracetamol/Tropisetron (Experimental)
  Interventions: Drug: Paracetamol; Drug: Tropisetron
- Saline (Placebo Comparator): Proband will receive Saline
  Interventions: Drug: Placebo
- Tropisetron (Active Comparator): Proband will receive Tropisetron alone
  Interventions: Drug: Tropisetron

INTERVENTIONS:
Drug: Paracetamol — Paracetamol 1 g i.v. once
  Arms: Paracetamol; Paracetamol/Tropisetron
Drug: Tropisetron — Tropisetron 5 mg i.v. once
  Arms: Paracetamol/Tropisetron; Tropisetron
Drug: Placebo — Saline
  Arms: Saline

SUMMARY:
1. Introduction

   Paracetamol, an analgesic prescribed daily, has been in use for more than 50 years. Surprisingly, its mode of action is still unclear. One postulated mechanism is the reinforcement of descending inhibitory pathways. A recent publication in a human pain model raises the question of whether or not Paracetamol acts according to a central serotonergic mechanism. Unfortunately, the chosen model was unable to differentiate between overall pain, secondary hyperalgesia and allodynia. In particular, secondary hyperalgesia and allodynia are central effects.

   The planned study will examine the central analgesic effects of paracetamol on allodynia and hyperalgesia by blocking the central effect by adding tropisetron. It will be based on an internationally accepted model for the initiation of secondary hyperalgesia, which was developed and tested by colleagues in Erlangen.
2. Study work plan

   This prospective, randomized, placebo-controlled, double-blinded, cross-over trial in 16 male volunteers will address pain ratings and the area of secondary hyperalgesia/allodynia in a human model of electrically evoked pain and compare four different treatment scenarios:
   * Paracetamol 1 g;
   * Paracetamol, 1 g and Tropisetron 5 mg;
   * Tropisetron, 5 mg; and
   * Saline.

   Each volunteer will be allocated to each scenario in a cross-over fashion. Four separate treatment trials, at least two weeks apart, will be performed. Each volunteer will be familiarized with the stimulation procedure prior to participation.
3. Ethical considerations

   Informed consent will be obtained from each volunteer. In addition, each volunteer will receive remuneration after participating in the study.

   Paracetamol is considered to be a very safe drug in healthy patients. Tropisetron, another safe medication, is routinely used in anaesthetic practice as an antiemetic drug. Headache, flush and liver parameter elevation are very rare side effects of minor importance in our daily clinical work as anaesthetists.

   This pain provoking procedure was developed at the University Erlangen Germany. It is a standardized method and has repeatedly received approval by research ethics committees internationally. Furthermore, the investigators applied this model to a recent study in Basel (cf your decision "study protocol 330/07;" unpublished data, analysis and writing in progress).
4. Patient number and timetable

   The investigators will examine 16 volunteers and expect the experimental component to last 3 months. The investigators plan to complete this study within one year.
5. Study importance

The mode of action of paracetamol remains unclear. The investigators think that this study will enable them to answer important questions concerning the action of paracetamol. The investigators hope that further understanding of this regularly prescribed drug will help us to better understand the complex mechanisms of pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* 20-35 years of age
* No known medical disorders
* BMI 18.5 - 39.9 (kg/m2)

Exclusion Criteria:

* Known drug allergies (paracetamol, tropisetron)
* Excessive consumption of tobacco (more than 10 cigarettes a day)
* Excessive consumption of tea or coffee (more than 5 cups a day)
* Recreational drug addiction
* Consumption of any medication on the trial days

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Pain | all 20 minutes up to 180 minutes after starting the experiment

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Ruppen, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital of Basel, Basel, Basel, Switzerland